## **SUMMARY OF CHANGES – Consent**

NCI Protocol #: 10450

**Local Protocol #:** 10450-36MTC **Protocol Version Date:** July 1, 2024

**Protocol Title:** A Phase Ib Trial of M3814 (Peposertib) in Combination with Lutetium 177 Dotatate for Well-Differentiated Somatostatin Receptor-Positive Gastroenteropancreatic

Neuroendocrine Tumors (GEP-NETs)

| # | Section | Comments |
|---|-------------------|-----------------------------------------------------|
| 1 | ICD-Global | The consent version date was updated. |
| 2 | Possible Side | Updated risks to match new CAEPR (Version 1.2, June |
| | Effects of | 12, 2024). |
| | <u>Peposertib</u> | |
| | (MSC2490484A) | Added New Risk: |
| | | Moved Risks: |

#### **Research Study Informed Consent Document**

**Study Title for Participants:** Testing the addition of an anti-cancer drug, Peposertib, to the usual radiation-based treatment (Lutetium Lu 177 Dotatate) for pancreatic neuroendocrine tumors

Official Study Title for Internet Search on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>: Protocol 10450, A Phase 1b Trial of M3814 (Peposertib) in Combination with Lutetium 177 Dotatate for Well-Differentiated Somatostatin Receptor-Positive Gastroenteropancreatic Neuroendocrine Tumors (GEP-NETs) (NCT: #NCT04750954)

## **Overview and Key Information**

## What am I being asked to do?

We are asking you to take part in a research study. This study has public funding from the National Cancer Institute (NCI), part of the National Institutes of Health (NIH) in the United States Department of Health and Human Services. We do research studies to try to answer questions about how to prevent, diagnose, and treat diseases like cancer.

We are asking you to take part in this research study because you have neuroendocrine tumors and your cancer is positive for somatostatin receptors.

## Taking part in this study is your choice.

You can choose to take part or you can choose not to take part in this study. You also can change your mind at any time. Whatever choice you make, you will not lose access to your medical care or give up any legal rights or benefits.

This document has important information to help you make your choice. Take time to read it. Talk to your doctor, family, or friends about the risks and benefits of taking part in the study. It's important that you have as much information as you need and that all your questions are answered. See the "Where can I get more information?" section for resources for more clinical trials and general cancer information.

## Why is this study being done?

This study is being done to answer the following question:

What is the highest dose of Peposertib in combination with Lutetium Lu 177 Dotatate that is safe and tolerable in patients with neuroendocrine tumors?

We are doing this study because we want to find out if this approach is better or worse than the usual approach for your neuroendocrine tumor. The usual approach is defined as care most people get for neuroendocrine tumors. There is evidence that the study drug, Peposertib, can make cancer more sensitive to the usual treatment, Lutetium Lu 177 Dotatate.

The combination of Peposertib and Lutetium Lu 177 Dotatate is not approved by the Food and Drug Administration (FDA) for any cancer.

This is the first time these drugs will be tested together in humans.

## What is the usual approach to my neuroendocrine tumor?

The usual approach for patients who are not in a study is treatment with Food and Drug Administration (FDA) approved drugs.

## What are my choices if I decide not to take part in this study?

- You may choose to have the usual approach described above.
- You may choose to take part in a different research study, if one is available.
- You may choose not to be treated for cancer.
- You may choose to only get comfort care to help relieve your symptoms and not get treated for your cancer.

## What will happen if I decide to take part in this study?

If you decide to take part in this study, you will get Peposertib and Lutetium Lu 177 Dotatate in combination for up to 32 weeks.

After you finish your study treatment, your doctor will continue to follow your condition every 4 months for 2 years from when you enrolled in this study or until your disease gets worse, and watch you for side effects with a procedure that uses a computer linked to an x-ray machine that takes detailed pictures of the areas inside your body. This is known as computer tomography (CT) scan. You will need to come to the clinic every 4 months during this follow-up period. This means you will keep seeing your doctor for up to 2 years after you enroll in this study.

## What are the risks and benefits of taking part in this study?

There are both risks and benefits to taking part in this study. It is important for you to think carefully about these as you make your decision.

#### Risks

We want to make sure you know about a few key risks right now. We give you more information in the "What risks can I expect from taking part in this study?" section.

If you choose to take part in this study, there is a risk that the study drugs may not be as good as the usual approach at shrinking or stabilizing your cancer.

There is also a risk that you could have side effects from the study drugs. These side effects may be worse and may be different than you would get with the usual approach for your cancer.

Some of the most common side effects that the study doctors know about are:



There may be some risks that the study doctors do not yet know about.

#### **Benefits**

There is some evidence from laboratory-based experiments that adding Peposertib to the usual approach can kill cancer cells, which might result in controlling cancer for longer than the usual approach alone. However, we do not know if this will happen in people. It is unlikely that adding Peposertib to the usual approach will help you live longer than the usual approach alone. This study may help the study doctors learn things that may help other people in the future.

## If I decide to take part in this study, can I stop later?

Yes, you can decide to stop taking part in the study at any time.

If you decide to stop, let your study doctor know as soon as possible. It's important that you stop safely. If you stop, you can decide if you want to keep letting the study doctor know how you are doing.

Your study doctor will tell you about new information or changes in the study that may affect your health or your willingness to continue in the study.

## Are there other reasons why I might stop being in the study?

Yes. The study doctor may take you off the study if:

- Your health changes and the study is no longer in your best interest.
- New information becomes available and the study is no longer in your best interest.
- You do not follow the study rules.
- For women: You become pregnant while on the study.
- The study is stopped by the Institutional Review Board (IRB), Food and Drug Administration (FDA), or study sponsor (NCI). The study sponsor is the organization who oversees the study.

It is important that you understand the information in the informed consent before making your decision. Please read, or have someone read to you, the rest of this document. If there is anything you don't understand, be sure to ask your study doctor or nurse.

## What is the purpose of this study?

The purpose of this study is to test the safety and tolerability of a drug called Peposertib in combination with Lutetium Lu 177 Dotatate. Peposertib has been tested in humans, but has not been tested in combination with Lutetium Lu 177 Dotatate in people with neuroendocrine tumors. There will be about 29 people taking part in this study.

## What are the study groups?

There are two parts in this study, a dose escalation part and a dose expansion part. Your doctor will tell you which part you are in.

In the dose escalation part of this study, different people will get different doses of the study drug Peposertib.

The first three people taking part in this study will get the starting dose of Peposertib. If the drug does not cause serious side effects, the next group of people in the study will get a higher dose. The study doctor will watch each group carefully as they increase the dose. The doses will continue to increase for every new group until people have serious side effects that require the dose to be lower. Once this dose is found, the dose escalation is stopped.

In the dose expansion part of this study, the highest dose with manageable side effects will be given to 14 more people. This will help study doctors better understand the side effects that may happen with this drug.

As of May 2023, the dose escalation part of the study has been completed and we have determined the dosages of Peposertib and Lutetium Lu 177 Dotatate to be used for the dose expansion part of the study.

Treatment schedule: You will get Lutetium Lu 177 Dotatate through a vein in your arm on the first day of each cycle. This will take approximately 30-40 minutes. You will take Peposertib by mouth \_\_\_\_\_\_\_. Your study doctor will tell you what dose to take. If you are in the dose escalation group, you will be asked to bring your morning dose of M3814 with you to the clinic on Days 9, 15, and 22 of Cycle 1. You will

be asked to fast (except for water) for 1 hour prior to dosing and for 1 hour after taking the oral dose of Peposertib. Peposertib tablets should not be crushed or opened. You should only take Peposertib and not take Peposertib until the bottle is empty. Peposertib should be stored at room temperature. Each cycle lasts 8 weeks. This study has 4 cycles. See the study calendar for more information.

You will not be able to get additional doses of the drug. This drug is not approved by the FDA for treatment of your disease.

Another way to find out what will happen to you during this study is to read the chart below. Start reading at the left side and read across to the right following the lines and arrows.

#### **Dose Escalation**



## What exams, tests, and procedures are involved in this study?

Before you begin the study, your doctor will review the results of your exams, tests, and procedures. This helps your doctor decide if it is safe for you to take part in the study. If you join the study, you will have more exams, tests, and procedures to closely monitor your safety and health. Most of these are included in the usual care you would get even if you were not in a study.

Listed below are exams, tests, and procedures that need to be done as part of this study to monitor your safety and health, but may not be included in the usual care. We will use them to carefully follow the effects of the study treatment, including preventing and managing side effects.

These exams, tests, and procedures to monitor your safety and health include:

- A computed tomography (CT) or magnetic resonance imaging (MRI) scan before you begin treatment, every 4 months during treatment, and when your disease gets worse.
- A gallium-68 dotatate positron emission tomography (PET)/CT scan before you begin treatment (or copper-64 dotatate PET/CT scan).
- Blood counts done before you begin study treatment, on Days 1, 9, 22, 29, and 43 of Cycle 1 of the study and then every 2-4 weeks afterward.
- Physical exams done monthly.
- For women able to have children, a pregnancy test before treatment begins. Short- and long-term safety data on fetuses exposed to Lutetium Lu 177 Dotatate are currently unknown. Pregnancy testing is being done to exclude pregnant patients from participating in this study.

Some exams, tests, and procedures are a necessary part of the research study, but would not be included in usual care. Listed below are procedures that will be done for research purposes only.

If you are in the dose escalation group, mandatory blood samples will be taken for the study. These required blood samples will be collected on Day 9 of Cycle 1 (9 times total over 8 hours) and one sample on Day 15 of Cycle 1 before you take your morning dose of Peposertib and one blood sample also on Day 22 of Cycle 1. These blood samples will help the researchers check the level of the study drug Peposertib in your blood at various time points (pharmacokinetics). You will not get any results of the blood tests.

A patient study calendar is attached at the end of this document. It shows how often these procedures will be done.

## What risks can I expect from taking part in this study?

#### **General Risks**

If you choose to take part in this study, there is a risk that the study drug may not be as good as the usual approach at shrinking or stabilizing your cancer.

You also may have the following discomforts:

- Spend more time in the hospital or doctor's office.
- Be asked sensitive or private questions about things you normally do not discuss.
- May not be able to take part in future studies.

The study drugs used in this study could be very harmful to an unborn or newborn baby. There may be some risks that doctors do not yet know about. It is very important that you check with your study doctor about what types of birth control or pregnancy prevention to use during the study and for 7 months after you have completed the study for women and for 4 months for men.

#### **Biopsy Risks**

Common side effects of a biopsy are a small amount of bleeding at the time of the procedure, bruising, and pain at the biopsy site. Pain can be treated with regular pain medications. Rarely, an infection can occur. You may sign a separate consent form for the study biopsy that describes the risks in more detail.

#### **Side Effect Risks**

The drugs used in this study may affect how different parts of your body work such as your liver, kidneys, heart, and blood. The study doctor will test your blood and let you know if changes occur that may affect your health.

There is also a risk that you could have other side effects from the study drug.

Here are important things to know about side effects:

- 1. The study doctors do not know who will or will not have side effects.
- 2. Some side effects may go away soon, some may last a long time, and some may never go away.
- 3. Some side effects may make it hard for you to have children.
- 4. Some side effects may be mild. Other side effects may be very serious and even result in death.

You can ask your study doctor questions about side effects at any time. Here are important ways to make side effects less of a problem:

- If you notice or feel anything different, tell your study doctor. He or she can check to see if it is a side effect.
- Your study doctor will work with you to treat your side effects.
- Your study doctor may adjust the study drugs to try to reduce side effects.

This study is looking at a combination of the usual drugs used to treat this type of cancer plus a study drug. This different combination of drugs may increase your side effects or may cause new side effects.

#### **Drug Risks**

The tables below show the most common and most serious side effects doctors know about. Keep in mind that there might be other side effects doctors do not yet know about. If important new side effects are found, the study doctor will discuss these with you.

#### Possible Side Effects of Peposertib (MSC2490484A)

(Table Version Date: June 12, 2024)



#### Possible Side Effects of Lutetium Lu 177 Dotatate

(Table Version Date: October 22, 2020)

#### OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving Lutetium Lu 177 dotatate, from 4 to 20 may have:

- Collection of immediate effects caused by a high dose of radiation, which includes loss of appetite
- Bruising, bleeding
- Infection, especially when white blood cell count is low

#### RARE, AND SERIOUS

In 100 people receiving Lutetium Lu 177 dotatate, 3 or fewer may have:

- Nausea, vomiting
- Cancer of bone marrow caused by chemotherapy
- Damage to the bone marrow (irreversible), which may cause infection, bleeding, and may require transfusions

#### **Additional Drug Risks**

The study drug could interact with other drugs and food including making one or more of your medications or the study medications work better or worse.

Your study

doctor will give you a Patient Drug Interactions handout and wallet card that lists the study treatment. Share this information with your family members, caregivers, other health care providers, and pharmacists.

Rarely, there are problems getting enough supplies of the study drug. If that happens, your doctor will talk with you about your options.

#### **Imaging Risks**

The gallium-68 (or copper-64) dotatate scan and 3D SPECT scans that you get in this study will expose you to low amounts of radiation. Every day, people are exposed to low levels of radiation that come from the sun and the environment around them. This type of radiation is called "background radiation." No one knows for sure whether exposure to these low amounts of radiation is harmful to your body.

The gallium-68 (or copper-64) dotatate scan and 3D SPECT scans that you get in this study will expose you to more radiation than you get from everyday background radiation. The amount of radiation from this scan is the same as 5 years of background radiation. Most of the time, this amount of extra radiation is not harmful to you. However, scientists believe that being exposed to too much radiation can cause harmful side effects. This could include getting a new cancer. We estimate that this could happen in about 1 out of every 1000 people who get a very large amount of extra radiation.

#### **Other Risks and Precautions**

Lutetium Lu 177 Dotatate, a beta- and gamma particle-emitting pharmaceutical, is a radioactive therapeutic agent. Though the external radiation exposure associated with Lutetium Lu 177 Dotatate is low, care must be used to keep body fluids from coming in contact with family members or caregivers. Your doctor will give you information on the good hygiene practices to follow to minimize radiation exposure from bodily fluids to household members and caregivers. Some of the precautions include using disposable gloves when wiping up blood, urine, stools, or vomit, or when handling stained clothes. Clothing soiled with Lutetium Lu 177 Dotatate or patient fecal matter or urine should be washed promptly and separately from other clothing. Use the same toilet each time you use the bathroom in your home, and if possible, use a different toilet than other members of your household. Sit down on the toilet to urinate to keep urine from splashing or spraying. Please follow these guidelines for at least 30 days after each Lutetium Lu 177 Dotatate treatment. Flush the toilet a few times after each use. Contact your health care team with questions you may have related to radiation exposure with Lutetium Lu 177 Dotatate.

## What are my responsibilities in this study?

If you choose to take part in this study you will need to:

- Keep your study appointments.
- Tell your doctor about:
  - o all medications and supplements you are taking
  - o any side effects
  - o any doctors' visits or hospital stays outside of this study
  - o if you have been or are currently in another research study.

• Write down in your medication diary when you take the study drug at home.

**For women:** Do not get pregnant while taking part in this study and for 7 months after the final dose of study medication. Do not breastfeed while taking part in this study and for 2.5 months after the final dose of study medication. **For men:** Do not father a baby while taking part in this study and use effective contraception for 4 months after the final dose of study medication. **For all:** Tell your study doctor right away if you think that you or your partner have become pregnant during the study or within 7 months after your last dose of Lutetium Lu 177 Dotatate.

## What are the costs of taking part in this study?

You and/or your insurance plan will need to pay for the costs of medical care you get as part of the study, just as you would if you were getting the usual care for your cancer. This includes:

- the costs of tests, exams, procedures, and drugs that you get during the study to monitor your safety, and prevent and treat side effects.
- the costs of getting Lutetium Lu 177 Dotatate ready and giving it to you.
- your insurance co-pays and deductibles.
- the gallium 68 dotatate scan (or copper-64 dotatate scan).
- the CT or MRI scans before you begin treatment, every 4 months during treatment, and when your disease gets worse.
- 24hr Urine Tests.
- EKG
- CT Scan.
- For women able to have children, a pregnancy test before you begin treatment.

Talk to your insurance provider and make sure that you understand what your insurance pays for and what it doesn't pay for if you take part in this clinical trial. Also, find out if you need approval from your plan before you can take part in the study.

Ask your doctor or nurse for help finding the right person to talk to if you are unsure which costs will be billed to you or your insurance provider.

You and/or your insurance provider will not have to pay for exams, tests, and procedures done for research purposes only or that are covered by the study. These include:

• The research blood draws on Day 9, Day 15 and Day 22 of Cycle 1, if you are in the dose escalation group.

You or your insurance provider will not have to pay for the Peposertib while you take part in this study.

Taking part in this study may mean that you need to make more visits to the clinic or hospital than if you were getting the usual approach to treat your cancer. You may:

- Have more travel costs.
- Need to take more time off work.
- Have other additional personal costs.

You will not be paid for taking part in this study. The research may lead to new tests, drugs, or other products for sale. If it does, you will not get any payment.

## What happens if I am injured because I took part in this study?

If you are injured as a result of taking part in this study and need medical treatment, please talk with your study doctor right away about your treatment options. The study sponsors will not pay for medical treatment for injury. Your insurance company may not be willing to pay for a study-related injury. Ask them if they will pay. If you do not have insurance, then you would need to pay for these medical costs.

If you feel this injury was caused by medical error on the part of the study doctors or others involved in the study, you have the legal right to seek payment, even though you are in a study. Agreeing to take part in this study does not mean you give up these rights.

## Who will see my medical information?

Your privacy is very important to us. The study doctors will make every effort to protect it. The study doctors have a privacy permit to help protect your records if there is a court case. However, some of your medical information may be given out if required by law. If this should happen, the study doctors will do their best to make sure that any information that goes out to others will not identify who you are.

Some of your health information, such as your response to cancer treatment, results of study tests, and medicines you took, will be kept by the study sponsor in a central research database. However, your name and contact information will not be put in the database. If information from this study is published or presented at scientific meetings, your name and other personal information will not be used.

There are organizations that may look at or receive copies of some of the information in your study records. Your health information in the research database also may be shared with these organizations. They must keep your information private, unless required by law to give it to another group.

Some of these organizations are:

- The study sponsor and any company supporting the study or the study agent now or in the future. This would include any organization helping the company with the study.
- The NCI Central IRB, which is a group of people who review the research with the goal of protecting the people who take part in the study.
- The FDA and the groups it works with to review research.
- The NCI and the groups it works with to review research.

• The Imaging and Radiation Oncology Core (IROC).

In addition to storing data in the study database, data from studies that are publicly funded may also be shared broadly for future research with protections for your privacy. The goal of this data sharing is to make more research possible that may improve people's health. Your study records may be stored and shared for future use in public databases. However, your name and other personal information will not be used.

Some types of future research may include looking at your information and information from other patients to see who had side effects across many studies or comparing new study data with older study data. However, right now we don't know what research may be done in the future using your information. This means that:

- You will not be asked if you agree to take part in the specific future research studies using your health information.
- You and your study doctor will not be told when or what type of research will be done.
- You will not get reports or other information about any research that is done using your information.

## Where can I get more information?

You may visit the NCI web site at http://cancer.gov/ for more information about studies or general information about cancer. You may also call the NCI Cancer Information Service to get the same information at: 1-800-4-CANCER (1-800-422-6237).

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

You can talk to the study doctor about any questions or concerns you have about this study or to report side effects or injuries. Contact the study doctor (\*insert name of study doctor[s]\*) at (\*insert telephone number, and email address if appropriate\*).

For questions about your rights while in this study, call the (\*insert name of organization or center\*) Institutional Review Board at (\*insert telephone number\*).

## Optional studies that you can choose to take part in

This part of the consent form is about optional studies that you can choose to take part in. They are separate from the main study described above. These optional studies will not benefit your health. The researchers leading these optional studies hope the results will help other people with your cancer in the future. The results will not be added to your medical records and you or your study doctor will not know the results.

Taking part in these optional studies is your choice. You can still take part in the main study even if you say "no" to any or all of these studies. There is no penalty for saying "no." You and

your insurance company will not be billed for these optional studies. If you sign up for, but cannot complete any of these studies for any reason, you can still take part in the main study.

Circle your choice of "yes" or "no" for each of the following studies.

#### Optional imaging study – research scan

If you are in the dose expansion group and choose to take part in this study, you will have seven scans at 1 hour, 4 hours, 1 day, 2 days, 3 days, 1 week, and 4 weeks following your first dose of Lutetium Lu 177 Dotatate. Researchers will use these scans to measure how Lutetium Lu 177 Dotatate moves through your body when used in combination with Peposertib. The scan will only be used for research and not to guide your medical care.

Please circle your answer: I choose to take part in the imaging study and will have the Lutetium Lu 177 Dotatate Dosimetry scans:

YES NO

## Optional sample collections for known laboratory studies and/or storage for possible future studies

Researchers are trying to learn more about cancer and other health problems using blood and tissue samples from people who take part in clinical trials. By studying these samples, researchers hope to find new ways to prevent, detect, treat, or cure diseases.

Some of these studies may be about how genes affect health and disease. Other studies may look at how genes affect a person's response to treatment. Genes carry information about traits that are found in you and your family. Examples of traits are the color of your eyes, having curly or straight hair, and certain health conditions that are passed down in families. Some of the studies may lead to new products, such as drugs or tests for diseases.

#### **Known future studies**

If you are in the dose expansion group and choose to take part in this optional study, researchers will collect your blood for research on evaluating the changes in your DNA and RNA that occur during treatment. Researchers will obtain genetic material (DNA and RNA) from both your tumor cells and your blood. Your DNA and RNA will be used for genomic sequencing, which is sequencing of all or part of your DNA. All your genetic information makes up your genome. Genomic sequencing is a test that records all or part of the pieces of DNA that are in your genes, piece by piece. This is usually done to look for changes in your genome that may cause health problems. The genomic sequencing will be done by an NCI-supported laboratory in Frederick, Maryland, known as the National Clinical Laboratory Network (NCLN) Genomics Laboratory at the Frederick National Laboratory for Cancer Research. The laboratory will compare the

genomic sequences from your tumor and blood cells to identify how they differ. The differences between genomic sequences of your tumor and blood cells may be important to understand why you did or did not respond to the treatment you received. Researchers hope to find potential "biomarkers" (changes present in tumor tissue that predict how patients with your type of cancer may respond to current or future treatments). This optional study may improve the ability to select future treatments or treatment combinations for others in the future. This optional study will not affect the cancer treatment or approach that you receive.

Neither you nor your study doctor will be informed when the genetic sequencing research will be done. You and your study doctor will not receive reports of these studies, as they are intended for research purposes only and cannot be used to plan treatment.

#### Unknown future studies

If you choose to take part in this optional study, a sample of your tumor tissue or blood samples left over from the genomic sequencing will be stored. Storing samples for future studies is called "biobanking." The biobank is being run by the Nationwide Children's Hospital in Columbus, Ohio, and is supported by the NCI. This is a publicly funded study. Samples from publicly funded studies are required to be shared as broadly as possible. However, we will protect your privacy. The goal of this is to make more research possible that may improve people's health.

The biobank is a public research resource. It has controlled access. This means that researchers who want to get samples and data from it must submit a specific research request. The request identifies who they are and what their planned research project is. Before getting the samples and data, the researchers must agree to keep the data private, only use it for their planned research project, and never use it to try to identify you.

Right now, we don't know what research may be done in the future using your tumor tissue and blood samples. This means that:

- You will not be asked if you agree to take part in the future research studies.
- You and your study doctor will not be told when or what type of research will be done.
- You will not get reports or other information about any research that is done using your samples.

#### What is involved in this optional sample collection?

If you agree to take part, here is what will happen next:

1. For patients in the dose escalation and dose expansion groups: About 2 teaspoons of blood will be collected from a vein in your arm before you begin study treatment, on Days 2 and 4 of cycle 1 (24 and 72 hours after your first dose of Lutetium Lu177 Dotatate at the time of the optional dosimetry scan), in the 4<sup>th</sup>, 8<sup>th</sup>, and 12<sup>th</sup> month after your first dose of Lutetium Lu177 Dotatate at the time of your CT scan to check your disease, and when your disease gets worse.

- 2. For patients in the dose expansion group only: A sample of tissue from a previous biopsy you had within 6 months before you begin the study will be sent to the biobank. If you do not have tissue available from a previous biopsy or if the biopsy was more than 6 months ago, samples of tissue will be collected from an optional extra biopsy before you begin study treatment. If you agree to have the sample of your tissue from a previous biopsy sent to the biobank or have the optional biopsy before you begin study treatment, the blood collection before you begin study treatment is mandatory.
- 3. Your samples will be stored in the biobank. There is no limit on the length of time we will keep your samples and research information. The samples will be kept until they are used for research or destroyed.
- 4. Researchers can only get samples from the biobank after their research has been approved by experts. Researchers will not be given your name or contact information.
- 5. Some of your genetic and health information may be placed in central databases for researchers to use. The databases will not include your name or contact information.

#### What are the risks in this optional sample collection?

- The most common risks related to drawing blood from your arm are brief pain and maybe a bruise.
- Generally, hospitals will keep some of your tissue. This tissue may be used to help treat your cancer in the future. There is a small risk that when this tissue sample is submitted to the biobank for this optional sample collection, your tissue could be used up.
- Your medical and genetic information is unique to you. There is a risk that someone
  outside of the research study could get access to your study records or trace information
  in a database back to you. They could use that information in a way that could harm you.
  Researchers believe the chance that someone could access and misuse your information is
  very small. However, the risk may increase in the future as people find new ways of
  tracing information.
- In some cases, this information could be used to make it harder for you to get or keep a job and get or keep health insurance. There are laws against the misuse of genetic information, but they may not give full protection. For more information about the laws that protect you, ask your study doctor or visit: https://www.genome.gov/10002328/

#### How will information about me be kept private?

Your privacy is very important to the study researchers and biobank. They will make every effort to protect it. Here are just a few of the steps they will take:

- 1. They will remove identifiers, such as your initials, from your sample and information. They will replace them with a code number. There will be a master list linking the code numbers to names, but they will keep it separate from the samples and information.
- 2. Researchers who study your samples and information will not know who you are. They also must agree that they will not try to find out who you are.
- 3. Your personal information will not be given to anyone unless it is required by law.

4. If research results are published, your name and other personal information will not be used.

#### What are the benefits to taking part in this optional sample collection?

You will not benefit from taking part.

The researchers, using the samples from you and others, might make discoveries that could help people in the future.

#### Are there any costs or payments to this optional sample collection?

There are no costs to you or your insurance. You will not be paid for taking part in this study. The research may lead to new tests, drugs, or other products for sale. If it does, you will not get any payment.

#### What if I change my mind about this optional sample collection?

If you decide you no longer want your samples to be used, you can call the study doctor, (\*insert name of study doctor for main trial\*), at (\*insert telephone number of study doctor for main trial\*), who will let the biobank know. Then, any sample that remains in the biobank will be destroyed or returned to your study doctor. This will not apply to any samples or related health information that have already been given to or used by researchers.

#### What if I have questions about this optional sample collection?

If you have questions about the use of your samples for research, contact the study doctor, (\*insert name of study doctor for main trial\*), at (\*insert telephone number of study doctor for main trial\*).

Please circle your answer below to show if you would or would not like to take part in each optional study:

#### Samples for known future studies:

I agree that my samples and related health information may be used for the laboratory studies described above.

YES NO

I agree that my study doctor, or someone on the study team, may contact me or my doctor to see if I wish to learn about results from these studies.

YES NO

## Samples for unknown future studies:

I agree that my samples and related health information may be kept in a biobank for use in future health research.

YES NO

This is the end of the section about optional studies.

## My signature agreeing to take part in the study

I have read this consent form or had it read to me. I have discussed it with the study doctor and my questions have been answered. I will be given a signed and dated copy of this form. I agree to take part in the main study. I also agree to take part in any additional studies where I circled "yes".

# Participant's signature

Signature of person(s) conducting the informed consent discussion

Date of signature

Date of signature

## **Patient Study Calendar**

| STUDY CALENDAR, Screening, Pre-Treatment and Cycle 1 | Screening | Pre-treatment | Day<br>1 | Day<br>2 | Day<br>4 | Day<br>9 | _ | cle 1 | Day 22 | Day 29 | Day 43 | Days<br>44-56 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Lutetium Lu 177 Dotatate | | | В | | | | | | | | | |
| | | | В | | | | | | | | | |
| Informed consent | X | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | |
| Medical history | X | | Х | | | | | | | X | | |
| Concurrent meds | X | | X | | | | | | | | | X |
| Physical exam | X | | X | | | | | | | X | | |
| Vital signs | X | | X | | | | | | | X | | |
| Height | X | | | | | | | | | | | |
| Weight | X | | Х | | | | | | | Х | | |
| Performance status | X | | Х | | | | | | | Х | | |
| CBC w/diff, plts | X | | X | | | X | X | X | X | X | X | |
| Comprehensive Chemistry Panel | X | | Х | | | X | X | Х | X | X | Х | |
| EKG (as indicated) | Х | | | | | | | | | | | |
| Gallium 68 (or Copper 64) Dotatate<br>PET/CT Scan | X | | | | | | | | | | | |
| Lutetium 177 Dosimetry | | | X | X | X | X | | | | X | | |
| Adverse Event evaluation | | | XX | | | | | | | | | |
| Radiologic evaluation | X | | Radiolo | ogic mea | suremen | ts should | l be perfo | rmed at | 4 montl | ns, 8 mont | ths, and 1 | 2 months |
| (CT/MRI Scan) | | | in the f | irst year | and then | every 4 | months u | ntil off | -study. | | | |
| Pregnancy test | X | | | | | | | | | | | |
| 24-Hour Urine 5HIAA | | | X | | | | | | | | | |
| PK blood sample collection<br>(mandatory; only in the dose<br>escalation cohort) | | | | | | Х | Х | | X | | | |
| Blood collection (Streck cfDNA) | | X | | | | | | | | | | |
| Whole Blood bio-banking (EDTA) | | X | Х | X | Х | | | | | | | |
| Archival Tumor tissue | | X | | | | | | | | | | |

| STUDY CALENDAR, Screening, Pre-Treatment | Screening | Pre-treatment | Cycle 1<br>(8-weeks) | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| and Cycle 1 | | | Day<br>1 | Day<br>2 | Day<br>4 | Day<br>9 | Day<br>15 | Day<br>21 | Day<br>22 | Day<br>29 | Day<br>43 | Days<br>44-56 |
| Research biopsy | | X | | | | | | | | | | |
| | | | C1<br>D1 | C1<br>D2 | C1<br>D4 | C1<br>D9 | C1<br>D15 | C1<br>D21 | C1<br>D22 | C1<br>D29 | C1<br>D43 | C1<br>D44-56 |

| STUDY CALENDAR, Cycles 2-4, Disease Progression & Follow-Up / Off-Treatment | | Cycle 2 (8-weeks) c | | | | Cycl<br>8-wee | | Cyc<br>3-we | ele 4<br>eks) | c | gression | Follow-up & Off-Treatment<br>Visits c, d, p, q | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| DAY(s) | 1 | 21 | 29 | 30-<br>56 | 1 | 21 | 29 | 30-<br>56 | 1 | 21 | 29 | 30-<br>56 | Disease Progression | Follow-up & Off<br>Visits c, d, p, q |
| Lutetium Lu 177 Dotatate | В | | | | В | | | | В | | | | | |
| Informed consent | | | | | | | | | | | | | | |
| Demographics | | | | | | | | | | | | | | |
| Medical history | X | | | | X | | | | X | | | | | |
| Concurrent meds | xx | | | | xx | | | | Х | | } | K | | |
| Physical exam | X | | X | | X | | X | | X | | X | | | X |
| Vital signs | X | | X | | X | | X | | X | | X | | | X |
| Height | | | | | | | | | | | | | | |
| Weight | X | | X | | X | | X | | X | | X | | | X |
| Performance status | X | | X | | X | | X | | X | | X | | | X |
| CBC w/diff, plts | X | | X | | X | | X | | X | | X | | | X |
| Comprehensive Chemistry Panel | | | X | | X | | X | | X | | X | | | Х |
| EKG (as indicated) | | | | | | | | | | | | | | |
| Gallium 68 (or Copper 64) Dotatate<br>PET/CT Scan | | | | | | | | | | | | | | |
| Lutetium 177 Dosimetry | | | | | | | | | | | | | | |
| Adverse Event evaluation | | xx | | | | ζ | X | | 2 | ζ | X | | | X |

| STUDY CALENDAR, Cycles 2-4, Disease Progression & Follow-Up / Off-Treatment | | | ycle 2<br>veeks | | ( | Cycl<br>8-wee | | (8 | Cyc<br>3-we | ele 4 | c | gression | Follow-up & Off -Treatment<br>Visits c, d, p, q | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| DAY(s) | 1 | 21 | 29 | 30-<br>56 | 1 | 21 | 29 | 30-<br>56 | 1 | 21 | 29 | 30-<br>56 | Disease Progression | Follow-up & C<br>Visits c, d, p, c |
| Radiologic evaluation (CT/MRI Scan) | | Radiologic measurements should be performed at 4 months, 8 months, and 12 months in the first year and then every 4 months until off-study. | | | | | | | | | | Х | | |
| Pregnancy test | | | | | | | | | | | | | | |
| 24-Hour Urine 5HIAA | | | | | Х | | | | | | | | | X |
| PK blood sample collection (mandatory) | | | | | | | | | | | | | | |
| Blood collection (Streck cfDNA) | | | | | | | | | | | | | X | |
| Whole Blood bio- banking (EDTA) | | | | | X | | | | | | | | X | Х |
| Archival Tumor tissue | | | | | | | | | | | | | | |
| Research biopsy | | | | | | | | | | | | | | |
| CYCLE | | | 2 | | | 3 | | | | 4 | | | | |

## STUDY CALENDAR Footnotes:

A: M3814 (peposertib): Dose as assigned . Cycle length = 8 weeks

B: Lutetium Lu 177 Dotatate: 200 mCi IV, Day 1 of each cycle for a total of 4 doses. Cycle length = 8 weeks.